CLINICAL TRIAL: NCT04692220
Title: Observatory of Drug-Related Problems: Impact of the Age and the Presence of Diabetes
Brief Title: Drug-Related Problems : Focus on Age and Diabetes
Acronym: DRP-AD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0667
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Adverse Drug Events
Keywords: Drug-Related Problems; Clinical Pharmacist; Elderly; Diabetes
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with an Adverse Drug Events or Drug-Related Problems: Patients with an Adverse Drug Events or Drug-Related Problems
  Interventions: Other: Detection of Adverse Drug Events or Drug-Related Problems
- Patients without an Adverse Drug Events or Drug-Related Problems: Patients without an Adverse Drug Events or Drug-Related Problems
  Interventions: Other: Detection of Adverse Drug Events or Drug-Related Problems

INTERVENTIONS:
Other: Detection of Adverse Drug Events or Drug-Related Problems — Detection of Adverse Drug Events or Drug-Related Problems

SUMMARY:
Drug-Related Problems (DRP) are a variety of events or circumstances that can interfere with the expected results of a treatment. They may be due to the drug itself, its association with other treatments, its incompatibility with the patient, its misuse... When these situations result in harm, they are referred to as adverse drug events (ADEs). DRP and particularly ADE represent a major public health problem in healthcare institutions because of their impact on morbidity and health costs.

DRPs are largely preventable and actions can be set up to detect and correct them. It is in this context that clinical pharmacy has expanded, with the development of new activities to help secure drug management. In our institution, the investigators have implemented several activities in different care services, including

* medication reconciliation,
* an ADE detection. These activities have interesting and encouraging results in terms of impact on the prevention of DRP. However, they can only be carried out on a limited number of patients, depending on the pharmaceutical resources available. The investigators therefore need tools to prioritize our activities on the most at-risk patients.

In this study, the investigators seek to identify DRP risk factors and develop DRP risk scores, with the objective to improve the detection and even prevention of DRP.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion criteria:

- Patients aged above 18 years old, admitted to the emergency department or hospital

Exclusion criteria:

* Patients presenting acute psychological disturbance
* Patients that did not agree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population was composed of patient admitted in emergency department or medical units of Montpellier University hospital.
Sampling Method: Non-Probability Sample
Enrollment: 27000 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
Variables associated with the presence of an Adverse Drug Events or Drug-Related Problems | 1 day
  Variables associated with the presence of an Adverse Drug Events or Drug-Related Problems

SECONDARY OUTCOMES:
Number and type of Adverse Drug Events and Drug-Related Problems | 1 day
  Number and type of Adverse Drug Events and Drug-Related Problems

CONTACTS AND LOCATIONS:
Overall Officials: Cyril BREUKER, PharmD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC